CLINICAL TRIAL: NCT03949907
Title: Early IntraVenous Administration of Nutritional Support (IVANS) in Metastatic Gastric, Cancer Patients at Nutritional Risk Undergoing First-line Chemotherapy
Brief Title: Early IntraVenous Administration of Nutritional Support
Acronym: IVANS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in anticancer treatment protocols which limit recruitment
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Director - Clinical Nutrition and Dietetics Unit, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190028466
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cancer of Stomach; GastroEsophageal Cancer
Keywords: Parenteral Nutrition (PN); Cancer
MeSH Terms: conditions — Stomach Neoplasms; Hyperphagia; Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional counseling alone (Other): Nutritional counseling consists of a personalized dietary prescription with regular consultation by a registered dietitian and telephone interviews, as well as of the use of oral nutritional supplements, when necessary.
  Interventions: Other: Nutritional counseling alone
- Supplemental parenteral nutrition plus nutritional counseling (Experimental): Patients will receive nutritional counseling in combination with systematic early supplemental home parenteral nutrition since diagnosis.
  Interventions: Other: Early supplemental parenteral nutrition plus nutritional counseling

INTERVENTIONS:
Other: Nutritional counseling alone — Nutritional counseling consists of a personalized dietary prescription (including sample meal plans and recipe suggestions) tailored on personal eating patterns and food preferences, in order to achieve estimated protein-calorie requirements and to take into account chewing and swallowing abilities. Regular consultation by a registered dietitian will be also provided every 10 days by means of face-to-face interviews (at scheduled follow-up visits - chemotherapy cycle) and telephone interviews (planned between chemotherapy cycles and as required by the patient). In the presence of significant reduction of normal food intake, the use of oral nutritional supplements will be also considered.
  In the presence of body weight loss >10% of the weight recorded at enrollment, patients allocated to this group group will be censored and treated according to current supportive care guidelines, including home parenteral nutrition.
  Arms: Nutritional counseling alone
Other: Early supplemental parenteral nutrition plus nutritional counseling — Patients will receive nutritional counseling in combination with systematic early supplemental home parenteral nutrition since diagnosis.
  Supplemental home parenteral nutrition will be prescribed, provided daily and adjusted throughout the study (approximately every 10 days, until the end of the scheduled first-line chemotherapy) according to estimated protein-calorie oral intakes, in order to satisfy estimated requirements. Home parenteral nutrition will be infused mainly during night hours, using multi-chamber bags containing olive oil-based lipid emulsions, when not contraindicated.
  Arms: Supplemental parenteral nutrition plus nutritional counseling

SUMMARY:
The present trial will be conducted to verify if early supplemental parenteral nutrition in combination with nutritional counseling improves survival and the feasibility of chemotherapy, in addition to nutritional status, body composition, functional status and quality of life in treatment-naïve patients with metastatic gastric cancer at nutritional risk undergoing first-line chemotherapy.

DETAILED DESCRIPTION:
Although it is known that nutritional support can improve clinical outcomes, the literature shows that only around 50% of cancer patients are able to satisfy estimated protein-calorie requirements. It is also emerging a strong correlation between nutritional status, particularly body composition, and adherence to active treatment. International guidelines suggest that parenteral nutrition (PN) is recommended in malnourished, hypophagic cancer patients suffering from gastrointestinal complications or with expected prolonged inadequate food intake, when enteral nutrition is not feasible. Although recent trials suggest that supplemental PN (SPN) could help to improve the nutritional status of malnourished cancer patients, there are no studies on the clinical effects of early SPN in cancer patients at nutritional risk receiving first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of metastatic gastric and gastroesophageal cancer;
* no previous chemotherapy for metastatic disease;
* indication for a first-line chemotherapy with a combination of 2 drugs including platinum derivatives (plus Trastuzumab if HER2+) to be used by investigator's choice within the framework of good clinical practice and in agreement with current Italian Association of Medical Oncology guidelines;
* measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST);
* presence of nutritional risk (Nutritional Risk Screening 2002 score ≥3);
* availability of permanent venous access (Port, Groshong, PICC);
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
* availability of a home parenteral nutrition service to continue nutritional plan as scheduled;
* signed informed consent.

Exclusion Criteria:

* age <18 years
* ECOG performance status >2
* indication to complete artificial nutrition support (totally compromised spontaneous food-intake)
* contraindication to parenteral nutrition (abnormal glucose and electrolytes control, hyper-triglyceridemia, impaired hemodynamic control and fluid retention)
* availability of jejunostomy for nutritional purposes
* ongoing home artificial nutrition
* unfeasible home parenteral nutrition for social/familial reasons
* absence of caregivers
* patients refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Combined endpoint - overall survival and weight maintenance | 12 months
  A combined endpoint consisting of overall and/or absence of unintentional weight loss >10% of the weight recorded at enrollment

SECONDARY OUTCOMES:
Overall survival | 12 months
  Overall survival
Treatment-related moderate-severe adverse events as assessed by CTCAE v4.0 | 4 months
  Difference in the incidence of grade >=3 toxicity, according to Common Terminology Criteria for Adverse Events [CTCAE v4.0]
Progression-Free Survival (PFS) | 12 months
  A progression-free survival rate at 12 months will be calculated, with patients categorized in a dichotomous manner as alive and progression-free or in progression or dead at 12 months.
Eligibility to second-line chemotherapy | 12 months
  The rate of patients eligible for second-line chemotherapy at 12 months will be calculated, with patients categorized in a dichotomous manner as alive and eligible or not eligible or dead at 12 months.
Total dose of chemotherapy administered | 4 months
  To be calculated as the percentage of chemotherapy dose administered with respect to the treatment plan
Objective response rate | 4 months
  Defined as a complete response or partial response that has been confirmed by a subsequent assessment no earlier than 2 months after the initial documentation. Response is assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Change in body weight | 12 months
  Change in body weight during the study (at 4 and 12 months)
Change in handgrip strength | 12 months
  Change in handgrip strength during the study (at 4 and 12 months)
Change in muscle mass | 12 months
  Change in muscle mass during the study (at 4 and 12 months) evaluated with computed tomography scan at the level of the third lumbar vertebra
Change in phase angle | 12 months
  Change in phase angle during the study (at 4 and 12 months) evaluated with bioimpedance vectorial analysis
Patients requiring unplanned hospitalization | 12 months
  The rate of patients requiring unplanned hospitalization (one or more) at 12 months will be calculated.
Change in self-perceived quality of life | 12 months
  Change in self-perceived quality of life during the study (at 4 and 12 months) as assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire version 3.0 [EORTC QLQ-C30]
Incidence of infections | 12 months
  The rate of incident infections in each group and the related difference will be calculated
Abnormal values in safety laboratory variables | 12 months
  The number of participants with abnormal values in safety laboratory variables will be calculated and compared between groups

OTHER OUTCOMES:
Serum levels of immunologic profiles | 1 months
  Levels of soluble effectors and immunoregulatory cells at 1 week and 1 month from the start of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Caccialanza, MD, Study Chair — Fondazione IRCCS Policlinico San Matteo; Emanuele Cereda, MD, PhD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo; Paolo Pedrazzoli, MD, Study Director — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Caccialanza R, Cereda E, Klersy C, Brugnatelli S, Borioli V, Ferrari A, Caraccia M, Lobascio F, Pagani A, Delfanti S, Aprile G, Reni M, Rimassa L, Melisi D, Cascinu S, Battistini L, Candiloro F, Pedrazzoli P. Early intravenous administration of nutritional support (IVANS) in metastatic gastric cancer patients at nutritional risk, undergoing first-line chemotherapy: study protocol of a pragmatic, randomized, multicenter, clinical trial. Ther Adv Med Oncol. 2020 Feb 22;12:1758835919890281. doi: 10.1177/1758835919890281. eCollection 2020. PMID 32127922